CLINICAL TRIAL: NCT07084610
Title: Metabolic Signatures Predictive of Response to Neoadjuvant Immunotherapy in Non-Small Cell Lung Cancer
Brief Title: Metabolic Biomarkers Predicting Response to Neoadjuvant Immunotherapy in Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital das Clínicas de Ribeirão Preto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 80521924.0.0000.5440; CAAE: 80521924.0.0000.5440 (Other: Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (HC-FMRP-USP))
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Platinum Compounds; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Single-arm, prospective, open-label study evaluating neoadjuvant nivolumab combined with chemotherapy in early-stage NSCLC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Nivolumab Plus Platinum-Based Chemotherapy (Experimental): Patients with resectable non-small cell lung cancer (NSCLC) clinical stage IB-IIIA (AJCC 8th edition) will receive two cycles of neoadjuvant nivolumab at 3 mg/kg combined with platinum-based doublet chemotherapy. Invasive mediastinal staging will be performed prior to neoadjuvant treatment. Following completion of systemic therapy, patients will undergo minimally invasive surgery (preferably robotic-assisted anatomical resection and mediastinal lymphadenectomy).
  Interventions: Drug: Nivolumab 3 mg/kg + platinum-based chemotherapy (2 cycles, neoadjuvant)

INTERVENTIONS:
Drug: Nivolumab 3 mg/kg + platinum-based chemotherapy (2 cycles, neoadjuvant) — Patients will receive neoadjuvant treatment with nivolumab (3 mg/kg, IV) combined with platinum-based chemotherapy (cisplatin 75 mg/m² or carboplatin AUC 5, plus pemetrexed 500 mg/m² for non-squamous or paclitaxel 175 mg/m² for squamous tumors) every 21 days for two cycles. All patients will undergo invasive mediastinal staging before treatment and will be treated with robotic-assisted anatomical lung resection and mediastinal lymphadenectomy after neoadjuvant therapy.
  Other Names: Neoadjuvant ICI + chemotherapy NSCLC

SUMMARY:
This study investigates metabolic glycolytic biomarkers obtained from radiological imaging (18F-FDG PET/CT), immunohistochemistry (IHC), and molecular analyses, and their association with response to neoadjuvant immunotherapy in early-stage non-small cell lung cancer (NSCLC).

Objective: To evaluate the relationship between glycolytic biomarkers measured by PET/CT (metabolic tumor volume and SUVmax), IHC markers (GLUT-1, Ki-67, PD-L1), and molecular oncogenic alterations, with the pathological response after two cycles of neoadjuvant nivolumab (3 mg/kg) combined with platinum-based chemotherapy in patients with early-stage NSCLC [stage IB (tumor ≥4 cm) to IIIA], negative for EGFR and ALK mutations.

Methods: This is a prospective, single-arm clinical study at a single institution, enrolling 30 patients. Baseline metabolic tumor volume (MTV) and SUVmax will be measured by PET/CT, while IHC markers and molecular profiling will be performed on pre-treatment biopsy samples. Patients will receive neoadjuvant treatment with nivolumab (3 mg/kg, IV) combined with platinum-based chemotherapy (cisplatin 75 mg/m² or carboplatin AUC 5, plus pemetrexed 500 mg/m² for non-squamous or paclitaxel 175 mg/m² for squamous tumors) every 21 days for two cycles. All patients will undergo invasive mediastinal staging before treatment and will be treated with robotic-assisted anatomical lung resection and mediastinal lymphadenectomy after neoadjuvant therapy. Primary outcomes include major pathological response (≤10% viable tumor cells) and immune profile characterization (IHC for CD8, CD4, FOXP3, PD-1, CD68, CD163). Secondary outcomes include event-free survival and treatment toxicity.

Standard of Care: Neoadjuvant chemotherapy regimens and PET/CT scans are part of the institutional standard of care for NSCLC patients.

Conclusion: The study aims to develop a practical diagnostic approach using metabolic glycolytic biomarkers to improve selection of patients likely to benefit from neoadjuvant immunotherapy. It is expected that patients with lower glycolytic activity will have higher rates of major pathological response after two cycles of neoadjuvant nivolumab (3 mg/kg) combined with chemotherapy. These findings may support a more cost-effective immunotherapy regimen for early-stage NSCLC.

DETAILED DESCRIPTION:
Introduction:

Metabolic reprogramming in cancer cells is an important feature that may impact response to immunotherapy. This study focuses on assessing glycolytic biomarkers through radiological (18F-FDG PET/CT), immunohistochemical (GLUT-1, Ki-67, PD-L1), and molecular analyses to better predict treatment outcomes in early-stage non-small cell lung cancer (NSCLC).

Study Design:

This is a prospective, single-arm, single-center clinical trial including 30 patients diagnosed with early-stage NSCLC (stages IB to IIIA) who are negative for EGFR and ALK mutations. All patients will receive two cycles of neoadjuvant nivolumab at 3 mg/kg combined with platinum-based chemotherapy (doublet regimen).

Procedures:

Before treatment, patients will undergo PET/CT scans to measure metabolic tumor volume (MTV) and maximum standardized uptake value (SUVmax). Tumor biopsies will be collected for immunohistochemistry and molecular profiling to evaluate markers such as GLUT-1, Ki-67, PD-L1, and oncogenic signaling pathways related to metabolism.

Endpoints:

Primary endpoints are major pathological response defined as ≤10% viable tumor cells in surgical specimens post-treatment, and immune microenvironment characterization through IHC markers (CD8, CD4, FOXP3, PD-1, CD68, CD163). Secondary endpoints include event-free survival, overall survival, and assessment of treatment-related toxicities.

Standard of Care:

Neoadjuvant chemotherapy and PET/CT imaging are part of routine clinical management for NSCLC at the institution.

Significance:

The study aims to provide a clinically feasible diagnostic tool to optimize patient selection for neoadjuvant immunotherapy, potentially enhancing efficacy and cost-effectiveness of treatment protocols in early-stage NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC), clinical stage IB to IIIA (according to AJCC 8th edition)
* Tumor deemed resectable by the multidisciplinary thoracic oncology team
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ and bone marrow function
* Ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* Prior systemic therapy, radiotherapy, or immunotherapy for lung cancer
* Known EGFR mutations or ALK rearrangements
* Active autoimmune disease requiring systemic therapy within the past 2 years
* Uncontrolled comorbidities or active infections
* Pregnant or breastfeeding women
* Contraindications to surgery or anesthesia
* Known history of other malignancies within the last 3 years, except for adequately treated basal or squamous cell skin cancer, or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) rate | At the time of surgery, approximately 6 to 8 weeks after the beginning of neoadjuvant treatment
  MPR will be defined as ≤10% of viable tumor cells in the resected surgical specimen, assessed by standardized pathological examination after lung resection.

CONTACTS AND LOCATIONS:
Overall Officials: Saulo B Silva, Associate Professor, MD, PhD, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (HC-FMRP-USP)
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (HC-FMRP-USP), Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to study outcomes (e.g., response to treatment, survival, toxicity) will be made available to researchers upon reasonable request, following publication of the main results. Data will be shared through institutional channels and upon approval by the principal investigator and ethics committee. Data will be available for a period of 5 years after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documentation will be available beginning 6 months after publication of the main results and will be accessible for up to 5 years.
Access Criteria: Qualified researchers may request access to de-identified individual participant data (IPD) and supporting documents (study protocol, SAP, ICF, CSR). Access will be granted upon reasonable request and after approval by the principal investigator and ethics committee. Requests must be made via email and include a research proposal and data use agreement.